CLINICAL TRIAL: NCT06937697
Title: Clinical Investigation of Hypersensitivity Reduction Efficacy on Colgate Dual Zinc Toothpaste Containing 5% Small Particle Size Silica (AC43) as Compared to Colgate MaxFresh Tea Toothpaste
Brief Title: Clinical of Hypersensitivity Reduction Efficacy on Two Toothpastes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-09-SEN-ZN-YPZ
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test 1 toothpaste (Experimental): Subjects will be instructed to brush their teeth with their assigned test dentifrice and toothbrush twice daily
  Interventions: Drug: Test toothpaste
- Control toothpaste (Active Comparator): Subjects will be instructed to brush their teeth with their assigned test dentifrice and toothbrush twice daily
  Interventions: Drug: Control toothpaste

INTERVENTIONS:
Drug: Test toothpaste — A commercially available fluoride toothpaste
  Arms: Test 1 toothpaste
Drug: Control toothpaste — A commercially available fluoride toothpaste
  Arms: Control toothpaste

SUMMARY:
To evaluate the clinical efficacy of a Dual Zinc Toothpast containing 5% small particle size silica (AC43) as compared to Colgate MaxFresh Tea Toothpaste on dentin hypersensitivity reduction after brushing two times daily (morning and evening) for a period of 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.
* Availability for the eight-week duration of the study.
* Two sensitive teeth, which must be anterior to the molars, and demonstrate cervical erosion/abrasion or gingival recession.
* Qualifying response to tactile stimuli (Yeaple probe) as defined by a score between 10-50 gms. of force.
* Qualifying response to the air blast stimuli as defined by a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale.
* Subjects need to satisfy the qualifying response to stimuli for both the parameters assessed (tactile or air) on two teeth to be entered into the study.
* Good general health with no known allergies to products being tested.
* Use of a non-desensitizing dentifrice for three months prior to entry into the study.
* Signed Informed Consent Form.

Exclusion Criteria:

* Gross oral pathology, chronic disease, or history of allergy to test products.
* Advanced periodontal disease or treatment for periodontal disease (including surgery) within the past twelve months.
* Sensitive teeth with a mobility greater than one.
* Teeth with extensive/defective restorations (including prosthetic crowns), suspected pulpitis, caries, cracked enamel, or used as abutments for removable partial dentures.
* Current use of anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs, or daily use of analgesics.
* Participation in a desensitizing dentifrice study or regular use of a desensitizing dentifrice within the past three months.
* Current participation in any other clinical study.
* Pregnant or lactating subjects.
* Allergies to oral care products, personal care consumer products, or their ingredients.
* Medical condition which prohibits not eating/drinking for 4 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
tactile sensitivity | baseline and 8 week measurement
  tactile stimulation is measured by the Yeaple Electronic Force Sensing Probe
air blast sensitivity | baseline and 8 week measurement
  air blast sensitivity is delivered by a standard dental unit syringe at a measured temperature of 19-21°C (70°F [± 3°F]) [sensitivity will be defined by a score of 2 or 3 on the Schiff Cold Air sensitivity scale Air Sensitivity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Deyu Hu, DDS, MS, Principal Investigator — West China Dental Institute of Chengdu
Locations (1):
- West China Dental Institute of Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No